CLINICAL TRIAL: NCT02975011
Title: Observational Study on the Effectiveness and Safety of Integrative Korean Medicine Treatment for Patients With Sciatica Due to Lumbar Stenosis: Multicenter, Prospective, Single Group Observational Study
Brief Title: Effectiveness and Safety of Korean Medicine for Lumbar Stenosis Patients With Sciatica
Status: Terminated | Type: Observational
Why Stopped: This study was prematurely terminated due to delayed patient enrollment.
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, Jinho Lee, Medical management director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2016-03
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Magnetic Resonance Imaging; Patient Satisfaction; Numeric Rating Scale
MeSH Terms: conditions — Spinal Stenosis; Patient Satisfaction | interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar stenosis group: Lumbar stenosis patients will be administered integrative Korean medicine treatment consisting of herbal medicine, Chuna manipulation, bee venom pharmacopuncture and pharmacopuncture, acupuncture, electroacupuncture, cupping, and other interventions, as needed.
  Interventions: Drug: Herbal medicine; Procedure: Chuna manipulation; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Other: Other intervention(s)

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine will be administered in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, Saposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycine max, Atractylodes japonica).
  Other Names: Traditional herbal medicine
Procedure: Chuna manipulation — Chuna is a Korean spinal manipulation that incorporates spinal manipulation techniques for joint mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manipulation will be administered to pelvic, lumbar, thoracic, and cervical vertebrae at the physician's discretion.
  Other Names: Chuna spinal manipulation
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture will be administered only after confirming a negative response to hypersensitivity skin test. Diluted bee venom (saline:bee venom ratio, 10,000:1) filtered for allergens will be injected at 4-5 acupoints proximal to the dysfunctional site at the physician's discretion. Each acupuncture point will be injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
  Other Names: Bee venom acupuncture
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Hyeopcheok (Huatuo Jiaji, EX B2), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Other: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary by the attending physician regardless of type or dose, and patterns of use will be investigated and recorded as an pragmatic clinical study.

SUMMARY:
A prospective study investigating the effectiveness and safety in lumbar stenosis patients receiving integrative Korean medicine treatment at 3 locations of Jaseng Hospital of Korean Medicine through assessment of pain, functional disability, and quality of life

DETAILED DESCRIPTION:
This is a prospective study to the aim of investigating the effectiveness and safety in patients with neurogenic claudication diagnosed as lumbar stenosis by lumbar MRI and receiving integrative Korean medicine treatment (herbal medicine, Chuna manipulation, bee venom pharmacopuncture and pharmacopuncture, acupuncture, electroacupuncture, and cupping) at 3 locations of Jaseng Hospital of Korean Medicine (Bucheon, Daejeon, Busan (Haeundae)) through assessment of pain, functional disability, and quality of life with 1-year follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiating leg pain with or without low back pain (LBP) (walking pain NRS ≥4)
* Patients with dural sac cross-sectional area (DSCA) of <100 mm2 or morphological grading ≥B as assessed on MRI
* Patients with clear neurogenic claudication symptoms (symptoms aggravated with walking, and alleviated upon resting in lumbar flexion position)
* Patients who have received surgery recommendation for lumbar spinal stenosis
* Patients with plans of receiving Korean medicine treatment for lumbar spinal stenosis for ≥2 months
* Patients who have agreed to study participation

Exclusion Criteria:

* Patients with vascular claudication
* Patients with other systemic diseases that may interfere with treatment effect or outcome interpretation
* Patients with soft tissue pathologies or pathologies of non-spinal origin that may cause LBP or radiating leg pain (e.g. spinal tumor, rheumatoid arthritis)
* Patients for whom acupuncture treatment may be inappropriate or unsafe (e.g. hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine intake, serious diabetes with risk of infection, severe cardiovascular diseases, or other conditions deemed unsuitable for acupuncture treatment)
* Pregnant patients or patients planning pregnancy
* Patients with serious psychological disorders
* Patients unable to fill out study participation consent form
* Subjects deemed unsuitable for study participation as assessed by the researchers

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lumbar stenosis patients with MRI results visiting and receiving treatment at 3 locations of Jaseng Hospital of Korean Medicine between November 2016 and March 2018
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Change in Numeric rating scale (NRS) of low back pain | Change from baseline to 3 months
  Change in low back pain intensity
Change in Numeric rating scale (NRS) of radiating leg pain | Change from baseline to 3 months
  Change in radiating leg pain intensity

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of low back pain | Baseline, 1, 2, 3, 6, 12 months
  Low back pain intensity for the past 3 days
Numeric rating scale (NRS) of radiating leg pain | Baseline, 1, 2, 3, 6, 12 months
  Radiating leg pain intensity for the past 3 days
Oswestry Disability Index (ODI) | Baseline, 1, 2, 3, 6, 12 months
  Functional disability questionnaire
EuroQol 5-dimensions 5-levels (EQ-5D-5L) | Baseline, 1, 2, 3, 6, 12 months
  Health-related quality of life questionnaire
Patient Global Impression of Change (PGIC) | 6, 12 months
  Global patient-reported outcome
Current medical service use | Baseline, 1, 2, 3, 6, 12 months
  Current use of medical services (type, frequency, period)
Pain-free walking time | Baseline, 1, 2, 3, 6, 12 months
  Average pain-free walking time for the past 3 days
Physical examination | Baseline, 1, 2, 3 months
  Lumbar physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Jinho Lee, KMD, Ph.D., Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No